CLINICAL TRIAL: NCT03499795
Title: A Phase 2, Open Label, Study of VGX-3100 Delivered Intramuscularly (IM) Followed by Electroporation (EP) for the Treatment of HPV-16 and/or HPV-18 Related Anal or Anal/Peri-Anal, High Grade Squamous Intraepithelial Lesion (HSIL), (AIN2, AIN3, PAIN2, PAIN3) in Individuals That Are Seronegative for Human Immunodeficiency Virus (HIV)-1/2
Brief Title: VGX-3100 Delivered Intramuscularly (IM) Followed by Electroporation (EP) for the Treatment of HPV-16 and/or HPV-18 Related Anal or Anal/Peri-Anal, High Grade Squamous Intraepithelial Lesion (HSIL) in Individuals Seronegative for Human Immunodeficiency Virus (HIV)-1/2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPV-203
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Anal Neoplasm
Keywords: High-grade squamous intraepithelial lesions (HSIL); Human papillomavirus (HPV); HPV-16; HPV-18; Anal intraepithelial neoplasia 2 (AIN2); Anal intraepithelial neoplasia 3 (AIN3); Peri-anal intraepithelial neoplasia 2 (PAIN2); Peri-anal intraepithelial neoplasia 3 (PAIN3)
MeSH Terms: conditions — Anus Neoplasms; Squamous Intraepithelial Lesions | interventions — VGX-3100

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VGX-3100 (Experimental): Adult participants who were HIV negative with histologically confirmed anal or anal/peri-anal HSIL associated with HPV-16 and/or 18, received four 6 mg doses of VGX-3100 as an IM injection on Day 0, Week 4, Week 12, and Week 40 followed immediately by EP using the CELLECTRA™ 5PSP device.
  Interventions: Biological: VGX-3100; Device: CELLECTRA™ 5PSP

INTERVENTIONS:
Biological: VGX-3100 — One milliliter (1 mL) VGX-3100 (deoxyribonucleic acid [DNA] plasmids encoding E6 and E7 proteins of HPV types 16 and 18) will be injected IM and delivered by EP using CELLECTRA™ 5PSP on Day 0, Week 4 and Week 12, and potentially Week 40.
Device: CELLECTRA™ 5PSP — IM injection of VGX-3100 is followed by EP with the CELLECTRA™ 5PSP device.

SUMMARY:
This is a phase 2, open-label efficacy study of VGX-3100 administered by intramuscular (IM) injection followed by electroporation (EP) in adult men and women who are human immunodeficiency virus (HIV) negative with histologically confirmed anal or anal/peri-anal high-grade squamous intraepithelial lesion (HSIL) associated with human papilloma virus (HPV)-16 and/or HPV-18. Approximately 24 participants will receive at least 3 doses of VGX-3100.

ELIGIBILITY:
Inclusion Criteria:

* Negative screening test for HIV-1/2 within 30 days of Dose 1;
* Confirmed anal or anal/peri-anal HPV-16/18 infection at Screening by polymerase chain reaction (PCR) from HSIL specimen;
* Anal tissue specimen/slides for diagnosis must be collected within 10 weeks of first dose of VGX-3100;
* At least one anal or anal/peri-anal (AIN2/3 and/or PAIN2/PAIN3) lesion that is histologically-confirmed as HSIL at Screening;
* Appropriate candidate for histology collection procedures (i.e. excision or biopsy) as judged by the Investigator;
* Female subjects must be post-menopausal, surgically sterile or agree to avoid pregnancy by continued abstinence or use of a contraceptive method with failure rate of less than 1% per year from Screening to one month after last dose of study medication (Week 12 or Week 40)
* Men who could father a child must agree to use at least one form of birth control during or continued abstinence from heterosexual intercourse prior to the study, for the duration of study participation and one month after last dose of study medication.
* Normal Screening electrocardiogram (ECG).

Exclusion Criteria:

* Untreated micro invasive or invasive cancer;
* Biopsy-proven Vaginal Intraepithelial Neoplasia (VAIN) and not undergoing medical care and/or treatment for VAIN;
* Biopsy-proven Vulvar Intraepithelial Neoplasia (VIN) and not undergoing medical care and/or treatment for VIN;
* Biopsy-proven Cervical Intraepithelial Neoplasia (CIN) 2/3 and not undergoing medical care and/or treatment for CIN;
* Biopsy-proven Penile Intraepithelial Neoplasia (PIN) and not undergoing medical care and/or treatment for PIN;
* Anal or anal/peri-anal HSIL that is not accessible for sampling by biopsy instrument;
* Intra-anal and/or peri-anal lesion(s) that cannot be fully visualized at Screening;
* Inability to have complete and satisfactory high resolution anoscopic exams (HRAs)
* Any treatment for anal or anal/peri-anal HSIL (e.g. surgery) within 4 weeks of Screening;
* Pregnant, breast feeding or considering becoming pregnant within one month following the last dose of study medication;
* Presence of any abnormal clinical laboratory values greater than Grade 1 per Common Toxicity Criteria for Adverse Events (CTCAE) version 4.03 within 45 days prior to Day 0 or less than Grade 1 but deemed clinically significant by the Investigator;
* Immunosuppression as a result of underlying illness or treatment;
* History of previous therapeutic HPV vaccination;
* Receipt of any non-study related non-live vaccine within 2 weeks of any VGX-3100 dose;
* Receipt of any non-study related live vaccine (e.g. measles vaccine) within 4 weeks of any VGX-3100 dose;
* Significant acute or chronic medical illness that could be negatively impacted by the electroporation treated as deemed by the Investigator;
* Current or history of clinically significant, medically unstable disease which, in the judgment of the investigator, would jeopardize the safety of the subject, interfere with study assessments or endpoint evaluation, or otherwise impact the validity of the study results;
* Prior major surgery within 4 weeks of Day 0;
* Participation in an interventional study with an investigational compound or device within 4 weeks of signing the ICF;
* Any illness or condition that in the opinion of the Investigator may affect the safety of the subject or the evaluation of any study endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (3):
- United States (2):
  - Howard Brown Health (HBH)-Sheridan, Chicago, Illinois
  - Laser Surgery Care, New York, New York
- Clinique de Recherche en Sante, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Canada and the United States from 15 May 2018 to 16 June 2020.
Pre-assignment Details: A total of 48 participants were screened out of which 23 were enrolled to receive study drug.
Groups:
- VGX-3100: Adult participants who were HIV negative with histologically confirmed anal or anal/peri-anal HSIL associated with HPV-16 and/or 18, received four 6 mg doses of VGX-3100 as an intramuscular (IM) injection on Day 0, Week 4, Week 12, and Week 40 followed immediately by electroporation (EP) using the CELLECTRA™ 5PSP device.
Period: Overall Study
Arm/Group | VGX-3100
Started | 23
Safety Population (Safety population included all participants who received at least 1 dose of VGX-3100+EP.) | 23
Modified Intent-to-treat (mITT) Population (mITT population included all participants who received at least 1 dose of VGX-3100+EP.) | 23
Completed | 21
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: mITT population included all participants who received at least 1 dose of VGX-3100+EP.
Arm/Group | VGX-3100
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 16
  Race: Other | 3
  Race: Black or African American | 2
  Race: Asian | 2
Region of Enrollment [Number; unit: participants]
  Canada | 4
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With no Histologic Evidence of Anal or Anal/Peri-Anal HSIL and no Evidence of HPV-16/18 at Week 36
Time Frame: Week 36
Population: mITT population included all participants who received at least 1 dose of VGX-3100+EP. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percentage of participants | 9.1 [1.6 to 25.9]
Statistical Analysis 1: Comparison: VGX-3100; Test type: Superiority; p = 0.8633, Clopper-Pearson; P-value was calculated based on the exact method of Clopper-Pearson and superiority was concluded if the one-sided p-value is <0.05

2. Secondary Outcome: Number of Participants With at Least One Local and Systemic Treatment-emergent Adverse Event (TEAE) During 7 Days Following Each Dose
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can include any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is any AE either reported for the first time or worsening of a pre-existing event after the first dose of study drug.
Time Frame: 7 days following each dose: Day 0 (Days 0 to 7), Week 4 (Days 22 to 28), Week 12 (Days 78 to 84), and Week 40 (Days 274 to 280)
Population: Safety population included all participants who received at least 1 dose of VGX-3100+EP.
Measure: Count of Participants; unit: Participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 23
Participants | 21

3. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can include any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From first injection up to Week 88
Population: Safety population included all participants who received at least 1 dose of VGX-3100+EP.
Measure: Count of Participants; unit: Participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 23
Participants | 23

4. Secondary Outcome: Percentage of Participants With no Evidence of Anal or Anal/Peri-Anal HSIL at Week 36
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percentage of participants | 13.6 [2.9 to 34.9]

5. Secondary Outcome: Percentage of Participants With no Evidence of HPV-16/18 From Intra-Anal and/or Peri-Anal Tissue by Type-Specific HPV Testing at Week 36
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percentage of participants | 45.5 [24.4 to 67.8]

6. Secondary Outcome: Percentage of Participants With no Evidence of HPV-16/18 From Intra-Anal Swab by Specific HPV Testing at Week 36
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percentage of participants | 31.8 [13.9 to 54.9]

7. Secondary Outcome: Percentage of Participants With no Evidence of Anal or Anal/Peri-Anal Low-Grade Squamous Intraepithelial Lesion (LSIL) or HSIL at Week 36
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percentage of participants | 9.1 [1.1 to 29.2]

8. Secondary Outcome: Percentage of Participants With no Progression of Anal or Anal/Peri-Anal HSIL to Carcinoma From Baseline to Week 36
Time Frame: From Baseline to Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percentage of participants | 100 [84.6 to 100]

9. Secondary Outcome: Percent Change From Baseline in the Number of Intra-Anal and/or Peri-Anal Lesions as Determined by the Investigator at Weeks 36, 64, and 88
Time Frame: From Baseline to Weeks 36, 64, and 88
Population: mITT population included all participants who received at least 1 dose of VGX-3100+EP. 'Overall number of participants analyzed' indicates the number of participants with data available for outcome measure analysis. 'Number analyzed' indicates the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percent change
  Percent Change From Baseline at Week 36 | -14.2 (41.93)
  Percent Change From Baseline at Week 64: number analyzed (Participants) | 21
  Percent Change From Baseline at Week 64 | -3.3 (37.91)
  Percent Change From Baseline at Week 88: number analyzed (Participants) | 21
  Percent Change From Baseline at Week 88 | -40.6 (46.77)

10. Secondary Outcome: Mean Change From Baseline in Frequency of HPV-16/17 E6/E7-specific CD8+/CD137+ Peripheral Blood Mononuclear Cells (PBMCs) That Were Perforin Positive at Week 15
Description: PBMCs were isolated from whole blood samples. The assessment of cellular immune activity occurred via the application Flow Cytometry for the purposes of performing a Lytic Granule Loading Assay. The Lytic Granule Loading assay examined cluster of differentiation (CD)8/CD137 cellular markers and Perforin (proteins involved in lytic degranulation and cytotoxic potential) intracellular marker. The frequency was presented as number of perforin-positive CD8 i.e., CD8+/ CD137+ PBMCs cells per million CD8+/ CD137+ PBMCs cells.
Time Frame: Baseline and Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells/million T cells + PBMCs
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
cells/million T cells + PBMCs | 4.491 (4.9686)

11. Secondary Outcome: Percentage of Participants With no Histologic Evidence of Anal or Anal/Peri-Anal HSIL or no Evidence of HPV-16/18 at Week 36
Time Frame: Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VGX-3100
Number analyzed (Participants) | 22
percentage of participants | 50.0 [28.2 to 71.8]

12. Other Pre Specified Outcome: Percent Change From Baseline in the Size of Peri-Anal Lesions as Determined by the Investigator at Weeks 36, 64, and 88
Time Frame: From Baseline to Weeks 36, 64, and 88
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From first injection up to Week 88
Description: Safety population included all participants who received at least 1 dose of VGX-3100+EP.
Arm/Group | VGX-3100
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 (N=23)
Ankle Fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VGX-3100 (N=23)
Nausea (Gastrointestinal disorders) | 10
Proctalgia (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Injection site pain (General disorders) | 20
Fatigue (General disorders) | 14
Injection site erythema (General disorders) | 7
Injection site pruritus (General disorders) | 6
Injection site bruising (General disorders) | 4
Injection site haemorrhage (General disorders) | 4
Injection site swelling (General disorders) | 4
Malaise (General disorders) | 4
Seasonal allergy (Immune system disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 8
Bronchitis (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 2
Arthropod bite (Injury, poisoning and procedural complications) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03499795/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03499795/SAP_001.pdf